CLINICAL TRIAL: NCT06748833
Title: An App Responding to Behaviour of People to Promote Mental Wellbeing in Anxious Youth
Acronym: SMILE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalhousie University (Other)
Responsible Party: Principal Investigator, Sandra Meier, Associate Professor, Dalhousie University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1026748_SMILE
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Anxiety; Sleep Problems
Keywords: anxiety; sleep problems; youths; mobile apps; mobile sensing; eHealth
MeSH Terms: conditions — Anxiety Disorders; Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SMILE Intervention Group (Experimental): The intervention group used the SMILE App, and the Predicting Risk and Outcomes of Social InTerActions (PROSIT) app, which is a mobile sensing app.
  Interventions: Behavioral: SMILE Intervention App
- Control Non-SMILE Intervention Group (No Intervention): Participants in the control group downloaded and used only the PROSIT app, they did not use the SMILE App.

INTERVENTIONS:
Behavioral: SMILE Intervention App — The SMILE app, an iOS and Android compatible smartphone app, is based on effective CBT-based treatment features to help patients manage anxiety symptomology. Access requires a unique login. The SMILE app utilizes three relaxation features: calm breathing, mindfulness meditation, and deep muscle relaxation; one cognitive feature, thought journaling and the challenging of thoughts; one self-monitoring technique; a positive imagery game; and a feature aimed to reduce avoidance behaviour through exposure. The app will be self-guided, with no additional human involvement needed. Participants will be instructed to actively engage with at least one of the app's major functions for a minimum of 3 minutes per day.
  Arms: SMILE Intervention Group

SUMMARY:
The goal of this clinical trial is to utilize mobile-sensing techniques to produce and test a simplified and personalized treatment app, Smile for Life (SMILE), for youth diagnosed with an anxiety disorder.

The main questions it aims to answer are:

1. What specific areas of difficulty (e.g., social interactions, physical activity/mobility, and sleep quality) are most impacted in youth with anxiety disorders, and how can a novel treatment app address these challenges?
2. Does the use of the novel treatment app lead to a measurable reduction in anxiety symptoms among youth, as assessed by the Screen for Child Anxiety Related Disorders (SCARED) survey, compared to a control group?

Researchers will compare the intervention to a control group (a group not given the SMILE app) to see if the intervention works to improve psychological functioning.

Participants will:

* Complete an online survey on emotional well-being and personality traits at the beginning and end of the one-month study, as well as at the 3-month follow-up. Participants will receive daily notifications asking participants to rate their social-emotional functioning. The app will then recommend a treatment plan and also ask participants to rate how helpful treatments were. Three months after the end of the study, participants will be asked to complete a follow-up assessment rating the app's usability.
* Participants in the intervention group will use a mobile app to practice cognitive behavioural therapy (CBT) treatment for their social-emotional issues.

DETAILED DESCRIPTION:
Background: The landscape of mental health treatment is expected to change due to the widespread use and availability of the Internet and mobile devices, as well as their increased capacity to deliver quality interventions. The development of treatment apps, such as the one investigated in the proposed study, will help to dismantle some of the barriers that prohibit youth from seeking or accessing treatment under the current health care model.

Smartphone interventions are particularly promising due to their ability to provide treatment exercises and monitor symptoms in situ (i.e., in real-time), immediately after or before pivotal events. A recent systematic review pointed out that some studies utilizing these digital interventions have high attrition rates; in some cases, rising as high as 70%. This is likely due to the fact that youth do not enjoy using digital health care systems that they perceive as impersonal and confusing to navigate.

Objective: Thus, the present study aims to determine which mobile-sensed daily life behaviours are indicative of anxiety problems by comparing the mobile- sensing profiles of youth with and without anxiety disorders as well as to evaluate the effectiveness of the novel treatment app on youth with anxiety disorders. The SMILE app incorporates Cognitive Behavioral Therapy (CBT) based treatment functions to help patients improve their mental health.

Method: Participants will be recruited and randomly allocated into the intervention and the control group. The study will measure anxiety, depression, drug and alcohol problems, and sleep problems before and after the one-month intervention period as psychological variables. Additionally, a 3-month follow-up will be the defining response of success for the SMILE app as participants will be asked to rate the app's ease of use, helpfulness, understandability, and if they would recommend the app to a friend.

Implications: If the intervention demonstrates effectiveness in reducing anxiety symptoms, it will undergo further testing to confirm its reliability and generalizability across diverse youth populations. Following these evaluations, the intervention will be integrated into the clinical care of youth with anxiety disorders, serving as both a stand-alone treatment option and a supplemental tool to complement existing therapeutic approaches, such as cognitive-behavioral therapy (CBT). This dual application will enable its use in various care settings, enhancing accessibility and providing tailored support to address the unique needs of individuals. Ultimately, the intervention aims to improve treatment outcomes, empower youth in managing their anxiety, and reduce the overall burden of anxiety disorders on mental health services.

The study will examine if a significant reduction of anxiety symptoms can be achieved in youth using the novel treatment app. We intend to recruit 120 participants with anxiety disorders between the ages of 12 and 21.

It is hypothesized that:

1. Youth with anxiety disorders will have fewer social interactions, be less physically active/mobile, and sleep worse, indicating areas in which these youth experience problems that the novel treatment app will need to focus on addressing using its features.
2. The effects of the novel treatment app will reduce youths' anxiety problems as measured by the SCARED survey compared to those in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read, write, and speak English
* Aged 12-21
* Regular access to and usage of a smartphone
* Score >25 on SCARED (25) (i.e., youth with anxiety disorders)

Exclusion Criteria:

* Other psychotherapy-based intervention
* Major medical illnesses which might impact participation (e.g., long periods of hospitalization)
* Youth who cannot provide informed consent (as this is a self-directed treatment program).

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 101 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Anxiety and sleep problems | One month
  Anxiety symptoms will be assessed using the 41-item SCARED questionnaire, where participants rate symptoms as not/hardly ever true (1), somewhat/sometimes true (2), or very/often true (3). Sleep problems will be assessed with the 7-item ISI, measuring difficulty falling/staying asleep and waking too early on a 5-point scale (0 = none, 4 = very severe). The ISI also evaluates sleep satisfaction, the noticeability of sleep issues, worry/distress about sleep, and their impact on daily functioning. Both tools will be administered pre- and post-intervention and at a three-month follow-up, providing comprehensive data on changes in anxiety and sleep problems over time. These measures will help determine the intervention's effectiveness in reducing anxiety and improving sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra M Meier, PhD, Principal Investigator — Dalhousie University
Locations (1):
- Dalhousie University, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
Participant data will be made available upon reasonable request to Dr. Sandra Meier (PI).